CLINICAL TRIAL: NCT02716090
Title: National Clinical Trial, Phase III, Monocentric, Randomized, Open, Controlled, Parallel Study to Assess the Non-inferiority of Dalap Duo® Product (0,1% Adapalene and 2,5% Benzoyl Peroxide Gel Cream) Compared to Epiduo® (0,1% Adapalene and 2,5% Benzoyl Peroxide Gel) in the Treatment of Acne Vulgaris in Population of Men and Women
Brief Title: Clinical Trial Phase III to Assess the Non-inferiority of Dalap Duo® Product Compared to Epiduo® in the Treatment of Acne Vulgaris
Acronym: Narciso
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to budget limitations, the company decided to withdraw this study.
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACH-DLP-03(01/13)
Record Dates: First submitted 2015-01-15; First posted 2016-03-23 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dalap Duo® (Experimental): 0.1% of adapalene and 2.5% and benzoyl peroxide gel cream. Apply the product on the areas affected by acne once a day in the evening for 84 days.
  Interventions: Drug: Adapalene and Benzoyl peroxide Dalap Duo®
- Epiduo® (Active Comparator): 0.1% of adapalene and 2.5% and benzoyl peroxide gel. Apply the product on the areas affected by acne once a day in the evening for 84 days.
  Interventions: Drug: Adapalene and Benzoyl peroxide Epiduo®

INTERVENTIONS:
Drug: Adapalene and Benzoyl peroxide Dalap Duo®
  Arms: Dalap Duo®
Drug: Adapalene and Benzoyl peroxide Epiduo®
  Arms: Epiduo®

SUMMARY:
This study evaluates the non-inferiority of the product Dalap Duo® compared to Epiduo® medicine to treat acne. Half of the participants will receive Dalap Duo®, while the other half will receive Epiduo®.

DETAILED DESCRIPTION:
The investigational product produced by Aché that will be evaluated in this trial is a cream gel, comprising 0.1% of adapalene 2.5% and benzoyl peroxide. It's a topical cream gel that is stored on a laminated tube containing 30 grams.

Of the 376 research participants with acne vulgaris participating in the study, 188 will be treated with the investigational product Cream Gel.

The duration of the participants in the study will be up to one hundred twenty-four days, contemplating screening visit, randomization visit, four follow-up visits, a final visit and a phone contact 30 days after final visit. Of the one hundred twenty and fourth days of the study period, the participants will be treated for eighty four days.

Regarding the control group, the active comparator is Epiduo®, manufactured by Galderma Laboratories, and its formulation is composed of 0.1% adapalene 2.5% and benzoyl peroxide. This is a topical gel stored in laminated tube with 30 grams.

Of the 376 research participants with acne vulgaris that will participate in the study, 188 will be treated with the active comparator Epiduo®.

The duration of the participants in the study will be up to one hundred twenty-four days, contemplating screening visit, randomization visit, four follow-up visits, a final visit and a phone contact 30 days after final visit. Of One hundred twenty and fourth days of the study period, the participants will be treated for eighty four days.

ELIGIBILITY:
Inclusion Criteria:

1. female or male Participant
2. Age older than or equal to 12 years;
3. 30-100 non-inflammatory facial lesions, except in the nose region (comedo closed and open comedo - degree 1) and 20 to 50 inflammatory facial lesions, except in the nose region (papule and pustule - degree 2);
4. Ability to understand and consent to participate in this clinical study, expressed by signing the consent form;
5. Search Participant willing to not use, for the entire period of the study drugs, cosmetics and / or treatments for acne, according to the investigator, that may influence the study results, such as, but not limited to, treatment with oral and topical retinoids.

Exclusion Criteria:

1. Any finding of clinical observation (clinical assessment / physical) that is interpreted by the investigator as a risk to safety or which may interfere with the effectiveness of the treatment and research of the participants in the clinical trial;
2. Any laboratory examination found that the investigator consider as safety risk or that may interfere with the effectiveness of the treatment and research of the participants in the clinical trial;
3. Known hypersensitivity to the drug components used during the study;
4. female participants with a history of polycystic ovary syndrome (Stein-Leventhal syndrome);
5. Women with positive result for urinary beta human chorionic gonadotropin or gestation period or breastfeeding;
6. Women in the reproductive age who do not agree to use acceptable contraception [oral contraceptives, injectable contraceptives, intrauterine device (IUD), hormonal implants, barrier methods, hormonal patch and tubal ligation]; other than surgically sterile (bilateral oophorectomy or hysterectomy) or sexual abstinence or who have not yet initiated sexual activity;
7. Person who has participated in clinical trial protocols in the last twelve (12) months, unless the investigator considers that there may be direct benefit to him/her;
8. Participant who has some kinship to the second degree or bond with employees or employees of Sponsor and Research Center;
9. Women in menopausal or postmenopausal period;
10. Any feature in the test areas (face) that according to the investigator may influence the results, for example, BUT NOT LIMITED TO moles, tattoos, scars, irritated skin, scratches, cuts and excess hair;
11. Participants diagnosed with Diabetes Mellitus after evaluation of the result of the test, defined as the presence of the classic symptoms of diabetes mellitus assessed the visit V-1 associated with the higher level of casual plasma glucose or equal to 200 mg / dL according to the American Diabetes Association (DIABETES CARE, VOLUME 33, SUPPLEMENT 1, JANUARY 2010);
12. Presence of dermatoses related to diabetes mellitus (plantar ulcer, necrobiosis lipoid, annular granuloma, dermatophytosis, deep mycoses, bacterial infections, opportunistic infections);
13. immune impairment;
14. Dermatological diseases in the test area (face): vitiligo, psoriasis, atopic dermatitis;
15. Participant using topical treatment for acne in the 15 days preceding the screening visit (V-1) or oral treatment for acne in the 30 days preceding the screening visit (V-1) or plan to use during the study period;
16. Participant with cyst or lump in the face region;
17. Use of medication and / or treatment contrary as described in item 11.2. of the Protocol;
18. Other diseases or medications, according to the investigator, that would interfere directly in the results of the study or jeopardize the health of the participant.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Reduction of total acne lesion | 84 days
  Percentage reduction of total acne lesion on the face other than the region of the nose by manual counting performed by the investigator.

SECONDARY OUTCOMES:
Reduction of number of inflammatory lesions | 07, 14, 28, 56 and 84 days
Reduction in non-inflammatory lesions | 07, 14, 28, 56 and 84 days
Improvement of acne through Global assessment of investigator | 07, 14, 28, 56 and 84 days
Efficiency perceived by participant | 84 days